CLINICAL TRIAL: NCT00994383
Title: A Single Dose, Three-Period, Three-Treatment, Six-Sequence, Three-Way Crossover Comparative Bioavailability Study of Morphine Sulfate Immediate Release Tablets and Solution and Controlled Release Capsules Under Steady-State Conditions.
Brief Title: Comparative Bioavailability Study of Morphine Sulfate Immediate Release and Controlled Release
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Elizabeth Ernst, Director, Drug Regulatory Affair and Medical Affairs, Roxane Laboratories, Inc.
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MORP-T30-PVFS-3
Record Dates: First submitted 2009-10-09; First posted 2009-10-14 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: morphine sulfate — morphine sulfate 30 mg tablet, morphine sulfate 15 mg tablet, morphine sulfate controlled release 120 mg
  Other Names: AVINZA

SUMMARY:
Characterize the steady-state pharmacokinetics of morphine after oral administration of Roxane Laboratories' morphine sulfate immediate release tablets and oral solution and to compare their pharmacokinetics to that of AVINZA.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening.

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C.
* Treatment with known enzyme altering drugs.
* History of allergic or adverse response to morphine sulfate or any comparable or similar product.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2007-01; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
bioequivalence determined by statistical comparison Cmax | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Fredrick A Bieberdorf, M.D., Principal Investigator — CEDRA Clinical Research
Locations (1):
- CEDRA Clinical Research, Austin, Texas, United States